CLINICAL TRIAL: NCT07159022
Title: High Flow Nasal Cannula and Mask Oxygenation in Patients With Visceral Obesity Undergoing Sedated Gastroscopy: A Randomized Controlled Trial.
Brief Title: High Flow Nasal Cannula and Mask Oxygenation in Patients With Visceral Obesity Undergoing Sedated Gastroscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B2025-212
Record Dates: First submitted 2025-08-27; First posted 2025-09-08 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: High Flow Nasal Cannula; Body Roundness Index

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Flow Nasal Cannula Oxygenation (Experimental): High Flow Nasal cannula is a system to deliver heated and humidified oxygen with an inspired oxygen fraction between 21 and 100% through large bore nasal cannula. The system delivers a flow up to 60 liters/min.
  Interventions: Procedure: High Flow Nasal Cannula Oxygenation
- Mask Oxygenation (Active Comparator): Conventional Oxygenation will be administered through mask
  Interventions: Procedure: Face Mask Oxygenation

INTERVENTIONS:
Procedure: High Flow Nasal Cannula Oxygenation — High Flow Nasal Cannula will be set at 60 liters per minute of air/oxygen admixture to reach a peripheral oxygen saturation equal or greater than 94%
  Arms: High Flow Nasal Cannula Oxygenation
Procedure: Face Mask Oxygenation — conventional oxygen therapy will be administered through common mask with a flow up to 6 Liters per minute
  Arms: Mask Oxygenation

SUMMARY:
During sedated gastroscopy, the insertion of the fiberscope and gastric distension required to perform the examination may induce respiratory depression, airway obstruction, and decreased chest wall compliance. Patients with obesity, especially visceral fat, have poor lung and chest wall compliance, lower lung capacity and functional residual capacity, and an unbalanced ventilation-to-perfusion ratio. Thus, obese patients are at a high risk of hypoxemia.

Increasing evidence supports the use of High-flow nasal cannula (HFNC) oxygenation in obese patients during sedated gastrointestinal endoscopy. Obesity, especially visceral obesity, is an established risk factor associated with all-cause mortality. Body roundness index (BRI) is a newer anthropometric measure associated with identification of high-risk individuals. Owing to the limited evidence, we designed this unblinded randomized controlled trial to assess whether HFNC, compared to standard mask oxygenation, improves oxygenation at the end of the procedure (primary endpoint) in patients with visceral obesity.

ELIGIBILITY:
Inclusion Criteria:

* ASA class ≤Ⅲ
* Visceral obesity（body mass index≥28 and BRI ≥5.46）
* Patients who will undergo sedated gastroscopy

Exclusion Criteria:

* Life-threatening heart disease or acute myocardial infarction within 6 weeks
* Presence of pneumothorax or pulmonary bullae, pulmonary embolism, pulmonary oedema
* Upper respiratory tract infection
* Presence of tracheostomy
* Nasal or nasopharyngeal diseases
* Coagulation disorders or a tendency of nose bleeding
* Pregnancy
* Recent (within 1 week) thoracic surgery
* Emergent procedure or surgery
* Allergy to drugs used during the procedure
* Unwillingness to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-31 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypoxia | From sedation with propofol to the end of the gastroscopy
  SpO2<90%

SECONDARY OUTCOMES:
Incidence of subclinical respiratory depression | From sedation with propofol to the end of the gastroscopy
  90%≤SpO2<95%
Severe hypoxia | From sedation with propofol to the end of the gastroscopy
  SpO2<75% for any duration or 75%≤SpO2<90% for >60 s
Serious cardiac events | Through gastroscopy completion, an average of 10-15 minutes
  Hypotension: Mean arterial pressure (MAP) < 65 mmHg; hypertension: MAP > 90 mmHg
Serious adverse respiratory events | Through gastroscopy completion, an average of 10-15 minutes
  Apnea, tracheospasm, larynx spasm

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospitla, Shanghai, China